CLINICAL TRIAL: NCT04073056
Title: Quadratus Lumborum II Block vs Conventional Therapy Alone For Laparoscopic Sleeve Gastrectomy
Brief Title: Efficacy Of Quadratus Lumborum II Block For Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ali Nima Shariat, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 18-1004
Record Dates: First submitted 2019-07-31; First posted 2019-08-28 (Actual); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Morbid Obesity; High BMI
Keywords: Sleeve gastrectomy; Quadratus lumborum block; Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum II Group (Active Comparator): The QL 2 group will receive 15 mL bupivacaine 0.25% on both sides for a total of 30 mL once the surgery is done but prior to extubation under ultrasound guidance.
  Interventions: Drug: Bupivacaine
- Conventional Therapy (Active Comparator): Conventional therapy consists of the injection of 30 mL of bupivacaine 0.25% directly into the incision sites by the surgeon at the end of the procedure.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine Hcl 0.25% Inj

SUMMARY:
The QL 2 block is a novel fascial plane block recently described by Blanco and colleagues in which local anesthetic is deposited adjacent to the antero-lateral aspect of the quadratus lumborum muscle. This results in posterior spread of local anesthetic through the middle layer of the thoraco-lumbar fascia, which theoretically communicates with the paravertebral space resulting in potentially longer-lasting and denser analgesia than wound infiltration. The QL 2 block derives from the TAP block, which is also a fascial plane block that is commonly used to treat pain following surgery involving the anterior abdominal wall. However, the QL block's more posterior location has recently been shown to provide a longer lasting and more profound analgesic effect than the TAP block, possibly by communicating with the paravertebral space. Although the TAP has been shown to be effective in a variety of surgical procedures involving an anterior abdominal wall incision including laparoscopic bariatric surgery the QL 2 block has until now, not been studied in the context of bariatric surgery.

DETAILED DESCRIPTION:
The QL 2 block is a novel fascial plane block recently described by Blanco and colleagues in which local anesthetic is deposited adjacent to the antero-lateral aspect of the quadratus lumborum muscle. This results in posterior spread of local anesthetic through the middle layer of the thoraco-lumbar fascia, which theoretically communicates with the paravertebral space resulting in potentially longer-lasting and denser analgesia than wound infiltration. Like the more commonly used transversus abdominis plane (TAP) block, the QL 2 block targets the anterior rami of T7-T12, ilioinguinal, iliohypogastric, and the lateral cutaneous branches of L1-L3. The QL 2 block derives from the TAP block, which is also a fascial plane block that is commonly used to treat pain following surgery involving the anterior abdominal wall. However, the QL block's more posterior location has recently been shown to provide a longer lasting and more profound analgesic effect than the TAP block, possibly by communicating with the paravertebral space. Although the TAP has been shown to be effective in a variety of surgical procedures involving an anterior abdominal wall incision including laparoscopic bariatric surgery the QL 2 block has until now, not been studied in the context of bariatric surgery. Conventional therapy has consisted of surgical infiltration of the incision ports with bupivacaine 0.25%. The study team proposes a study to compare the analgesic effects of the QL 2 block with conventional therapy, consisting of surgical wound infiltration, for postoperative analgesia following laparoscopic gastric sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo laparoscopic gastric sleeve gastrectomy
* 18-65 years of age
* BMI> 35 kg/m2.

Exclusion Criteria:

* Contraindications to administration of local anesthesia (e.g. local anesthetic allergy)
* Contraindication/allergy to acetaminophen or ketorolac
* History of substance abuse or chronic opioid use
* Coagulopathy
* Patients receiving systemic anticoagulation
* Local infection
* ASA 4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali N Shariat, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai St. Lukes Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King WC, Chen JY, Belle SH, Courcoulas AP, Dakin GF, Flum DR, Hinojosa MW, Kalarchian MA, Mitchell JE, Pories WJ, Spaniolas K, Wolfe BM, Yanovski SZ, Engel SG, Steffen KJ. Use of prescribed opioids before and after bariatric surgery: prospective evidence from a U.S. multicenter cohort study. Surg Obes Relat Dis. 2017 Aug;13(8):1337-1346. doi: 10.1016/j.soard.2017.04.003. Epub 2017 Apr 7. PMID 28579202
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Background] Albrecht E, Kirkham KR, Endersby RV, Chan VW, Jackson T, Okrainec A, Penner T, Jin R, Brull R. Ultrasound-guided transversus abdominis plane (TAP) block for laparoscopic gastric-bypass surgery: a prospective randomized controlled double-blinded trial. Obes Surg. 2013 Aug;23(8):1309-14. doi: 10.1007/s11695-013-0958-3. PMID 23591549
- See also: King WC, Chen J-Y, Belle SH, et al.; Use of Prescribed Opioids Before and After Bariatric Surgery: Prospective Evidence from a U.S. Multicenter Cohort Study Surg Obes Relat Dis 2017; 13: 1337-1346. — https://www.ncbi.nlm.nih.gov/pubmed/28579202
- See also: Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarian Delivery. Reg Anesth Pain Med 2016; 41: 757-762. — https://www.ncbi.nlm.nih.gov/pubmed/27755488
- See also: Albrecht E, Kirkham KR, Endersby RVW, et al. Ultrasound-Guided Transversus Abdominis Plane (TAP) Block for Laparoscopic Gastric-Bypass Surgery: a Prospective Randomized Controlled Double-Blinded Trial. Obes Surg 2013; 23: 1309-1314. — https://www.ncbi.nlm.nih.gov/pubmed/23591549

RESULTS

PARTICIPANT FLOW:
Groups:
- Quadratus Lumborum II Group: The QL 2 group received 15 mL bupivacaine 0.25% on both sides for a total of 30 mL once the surgery is done but prior to extubation under ultrasound guidance.
  Bupivacaine: Bupivacaine Hcl 0.25% Inj
Period: Overall Study
Arm/Group | Quadratus Lumborum II Group | Conventional Therapy
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Therapy | Quadratus Lumborum II Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (11.3) | 37.4 (9.84) | 38.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 42.9 (5.50) | 43.3 (7.46) | 43.1 (6.47)
Existence of preexisting pain [Count of Participants; unit: Participants] | 5 | 5 | 10
Pre Non-analgesic Meds [Count of Participants; unit: Participants] | 12 | 13 | 25
Pre Analgesic Meds [Count of Participants; unit: Participants] | 2 | 1 | 3
Recreational drug use [Count of Participants; unit: Participants] | 4 | 1 | 5
Preop Systolic Blood Pressure (BP) [Mean (Standard Deviation); unit: mmHg] | 125 (9.51) | 127 (14.2) | 126 (12.0)
Preop Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 80.0 (8.19) | 79.5 (8.24) | 79.7 (8.11)
Preop Mean Arterial Pressure (MAP) [Mean (Standard Deviation); unit: mmHg] | 90.2 (22.4) | 95.2 (9.25) | 92.7 (17.1)
Preop Heart Rate (HR) [Mean (Standard Deviation); unit: beats per minute] | 87.4 (12.0) | 84.3 (15.7) | 85.8 (13.9)
Preop Respiratory Rate (RR) [Mean (Standard Deviation); unit: breaths per minute] | 16.3 (1.14) | 17.9 (2.66) | 17.1 (2.15)
Preop Oxygen Saturation (SpO2) [Mean (Standard Deviation); unit: percent] — Oxygen saturation measured by pulse oximetry
  percent | 98.5 (0.820) | 98.0 (1.34) | 98.3 (1.12)

OUTCOME MEASURES:

1. Primary Outcome: The Amount of Opioid Consumption During and After Procedure
Description: The amount of opioid consumption (in mg IV morphine equivalents) during and after procedure (100mcg fentanyl= 10mg morphine) (1.5mg dilaudid=10mg morphine)
Time Frame: Intraop, Postop 1hr, Postop 2hr, POD0, POD1, and POD2
Population: Post Anesthesia Care Unity (PACU) hr 2 - one participant from each group was ready for discharge from the PACU prior to the 2nd hour.
  Postop Day (POD) 2 - two participants from each group could not be reached by phone.
Measure: Mean (Standard Deviation); unit: mg IV morphine equivalents
Groups:
- Quadratus Lumborum II Group: The QL 2 group received 15 mL bupivacaine 0.25% on both sides for a total of 30 mL once the surgery is done but prior to extubation under ultrasound guidance.
Arm/Group | Conventional Therapy | Quadratus Lumborum II Group
Number analyzed (Participants) | 20 | 20
mg IV morphine equivalents
  Intraop | 26.3 (12.4) | 27.1 (11.9)
  POQ1 - PACU hour 1 | 5.49 (3.49) | 5.52 (3.64)
  POQ2 - PACU hour 2: number analyzed (Participants) | 19 | 19
  POQ2 - PACU hour 2 | 2.80 (1.66) | 1.68 (2.10)
  POD 0 | 4.14 (5.12) | 2.53 (3.16)
  POD1 | 3.13 (4.72) | 2.75 (3.52)
  POD2: number analyzed (Participants) | 18 | 18
  POD2 | 0.938 (1.46) | 0.750 (1.43)

2. Secondary Outcome: VAS Pain Scores
Description: Visual analogue scale - total score from 0 to 10, with higher score indicating more pain
Time Frame: Intraop, Postop 1hr, Postop 2hr, POD0, POD1, and POD2
Population: PACU hr 2 - one participant from each group was ready for discharge from the PACU prior to the 2nd hour.
  POD 2 - two participants from each group could not be reached by phone.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Therapy | Quadratus Lumborum II Group
Number analyzed (Participants) | 20 | 20
score on a scale
  POQ1 - PACU hour 1 | 6.60 (2.11) | 6.15 (1.95)
  POQ2 - PACU hour 2: number analyzed (Participants) | 19 | 19
  POQ2 - PACU hour 2 | 4.37 (2.27) | 3.11 (1.59)
  POD 0 | 5.85 (2.89) | 4.80 (2.33)
  POD1 | 6.20 (2.71) | 4.05 (1.96)
  POD2: number analyzed (Participants) | 18 | 18
  POD2 | 5.00 (2.57) | 3.28 (1.87)

3. Secondary Outcome: Respiratory Rate
Description: Respiratory rate in breaths per minute
Time Frame: 1 hour post op
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Conventional Therapy | Quadratus Lumborum II Group
Number analyzed (Participants) | 20 | 20
breaths per minute | 22.5 (2.72) | 17.0 (4.80)

4. Secondary Outcome: Heart Rate
Description: Heart rate in beats per minute
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Conventional Therapy | Quadratus Lumborum II Group
Number analyzed (Participants) | 20 | 20
beats per minute | 85.3 (14.0) | 7.3 (12.5)

5. Secondary Outcome: Blood Pressure
Description: Both systolic and diastolic pressures
Time Frame: 1 hour after surgery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Conventional Therapy | Quadratus Lumborum II Group
Number analyzed (Participants) | 20 | 20
mmHg
  Systolic pressure | 134 (11.9) | 136 (15.9)
  Diastolic | 80.1 (11.6) | 83.0 (10.8)

6. Secondary Outcome: Time to First Dose of Analgesic Request
Description: Time until first analgesic request in minutes
Time Frame: up to 60 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Conventional Therapy | Quadratus Lumborum II Group
Number analyzed (Participants) | 20 | 20
minutes | 34.0 (23.9) | 28.1 (18.4)

7. Secondary Outcome: PACU Length of Stay
Description: Post anesthesia care unit (PACU) length of stay in hours
Time Frame: average 2 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Conventional Therapy | Quadratus Lumborum II Group
Number analyzed (Participants) | 20 | 20
hours | 2.18 (0.572) | 1.95 (0.822)

8. Secondary Outcome: Number of Participants With Pain
Description: Number of participants with somatic or visceral pain.
Time Frame: Up to 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Therapy | Quadratus Lumborum II Group
Number analyzed (Participants) | 20 | 20
Participants
  Somatic pain | 3 | 2
  Visceral pain | 18 | 18

9. Secondary Outcome: Number of Participants With Nausea
Description: Number of participants with nausea
Time Frame: the first 48 hours after the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Therapy | Quadratus Lumborum II Group
Number analyzed (Participants) | 20 | 20
Participants
  POQ2 | 12 | 7
  POD1 | 8 | 6
  POD2 | 4 | 2

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Quadratus Lumborum II Group | Conventional Therapy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT04073056/Prot_000.pdf
  • Informed Consent Form (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT04073056/ICF_001.pdf